CLINICAL TRIAL: NCT03684772
Title: A Phase 2, Randomized, Double Blind, Vehicle Controlled, Parallel Group Study to Explore the Efficacy, Pharmacodynamics and Safety of Topical Ionic Contra-Viral Therapy (ICVT) Comprised of Digoxin and Furosemide in Actinic Keratosis
Brief Title: Topical Ionic Contra-Viral Therapy in Actinic Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS003-CO-PR-004
Record Dates: First submitted 2018-08-23; First posted 2018-09-26 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICVT (Experimental): Digoxin and Furosemide (0.125%)
  Interventions: Drug: ICVT Topical Gel
- Furosemide (Experimental): Furosemide (0.125%)
  Interventions: Drug: Furosemide Topical Gel
- Digoxin (Experimental): Digoxin (0.125%)
  Interventions: Drug: Digoxin Topical Gel
- Placebo (Placebo Comparator): Vehicle Gel
  Interventions: Drug: Vehicle Topical Gel

INTERVENTIONS:
Drug: ICVT Topical Gel — Digoxin and Furosemide (0.125%)
  Arms: ICVT
Drug: Furosemide Topical Gel — Furosemide (0.125%)
  Arms: Furosemide
Drug: Digoxin Topical Gel — Digoxin (0.125%)
  Arms: Digoxin
Drug: Vehicle Topical Gel — Vehicle Gel
  Arms: Placebo

SUMMARY:
To explore the pharmacodynamics and evaluate safety, tolerability and clinical efficacy of ICVT comprised of digoxin and furosemide (dual agent), digoxin (single agent), furosemide (single agent) in patients with AK.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects 18 years or older with verified condition of general good health (with exception of AK)
* Confirmed clinical AK diagnosis by dermatologist
* Subjects must have at least 2 facial fields of at least 25 cm² (but preferably >35 cm²) present at screening and baseline visit where more than 2 AK lesions are visible in each field (preferably the forehead, temple or cheek)
* Subjects must be able to participate and willing to give written informed consent and to comply with the study restrictions
* Subjects must be able to communicate well with the investigator in Dutch
* Subjects willing to refrain from using other topical products in the treatment area, or prohibited medication for the duration of the study
* Subjects must be willing to limit sun exposure of the involved skin to the extent vocationally possible
* Subjects and their partners of childbearing potential must use effective contraception, for the duration of the study and for 3 months after the last dose.

Exclusion Criteria:

* Have used or received any treatment for AK in the treatment area within 28 days prior to enrollment (including topical medications, immunosuppressive or immunomodulating agents, phototherapy, oral retinoids, or other therapies for AKs)
* Have any current pathologically relevant skin conditions in the field area other than AK (e.g. squamous cell carcinoma or basal cell carcinoma).
* Have a known hypersensitivity to any of the investigational product ingredients, including digoxin and furosemide.
* Current use of systemic digoxin or furosemide.
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year
* Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening or intention to donate blood or blood products during the study.
* If a woman of childbearing potential, pregnant, or breast-feeding, or planning to become pregnant during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Complete clinical clearance (CCC) per field | Day 42
Change in AK-FAS (AK field assessment scale) | Day 42
  AK Grade 0-IV, the higher the number the more % area covered by AK
Investigator global score (IGS) of each field | Day 126
  This is a 7 point scale from -2 (significantly worse) to +4 (completely cured), higher values represent a better outcome
Evolution of one assigned target lesion in the field, assessed by dermoscopy | Day 126
  assessing erythema, scaling, pigmentation, and follicular plug
Field morphology | Day 126
  Change in lesion count per field
Standardized photography with Canfield VISIA or 2D photography and with Antera 3D camera | Day 126
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: IFN-a. IFN-g, Ki-67
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: IFN-g
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: Ki-67
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: p53
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: MCM7(minichromosome maintenance protein 7)
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker:putrescene
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: spermidine
Biopsy biomarker | Day 126
  Analysis will be prerformed for the following biomarker: beta HPV types 5,8,15,20,24,38
Skin swab markers | Day 126
  Swab analysis will be performed for beta HPV types 5,8,15,20,24,38.

SECONDARY OUTCOMES:
Adverse events collected throughout the study | Day 126
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: Heart Rate (bpm
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: PR
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: QRS
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: QT
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: QTcB
12-Lead ECGs performed at Screening and End of Study | Day 126
  The following component will be assessed: QTcF
Vital Signs performed at Screening and End of Study | Day 42
  The following will be assessed: Pulse Rate (bpm)
Vital Signs performed at Screening and End of Study | Day 42
  The following will be assessed: Systolic blood pressure (mmHg)
Vital Signs performed at Screening and End of Study | Day 42
  The following will be assessed: Diastolic blood pressure (mmHg)
Vital Signs performed at Screening and End of Study | Day 42
  The following will be assessed: Temperature ( ̊ C)
Patient diary on treatment application compliance, local tolerance and selfies photo | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands